CLINICAL TRIAL: NCT05052801
Title: A Randomized, Multi-center, Double-blind, Placebo-controlled Phase 3 Study of Bemarituzumab Plus Chemotherapy Versus Placebo Plus Chemotherapy in Subjects With Previously Untreated Advanced Gastric or Gastroesophageal Junction Cancer With FGFR2b Overexpression
Brief Title: Bemarituzumab or Placebo Plus Chemotherapy in Gastric Cancers With Fibroblast Growth Factor Receptor 2b (FGFR2b) Overexpression
Acronym: FORTITUDE-101
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Collaborators: Zai Lab (China only) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20210096; 2023-505457-40 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2021-09-13; First posted 2021-09-22 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Gastric Cancer; Gastroesophageal Junction Adenocarcinoma
Keywords: Gastric Cancer; Gastroesophageal Junction Adenocarcinoma; Bemarituzumab; FGFR2b Overexpression
MeSH Terms: conditions — Stomach Neoplasms | interventions — bemarituzumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Bemarituzumab with mFOLFOX6 (Experimental)
  Interventions: Drug: Bemarituzumab; Drug: mFOLFOX6
- Placebo with mFOLFOX6 (Active Comparator)
  Interventions: Drug: mFOLFOX6; Drug: Placebo

INTERVENTIONS:
Drug: Bemarituzumab — Intravenous (IV) infusion
  Arms: Bemarituzumab with mFOLFOX6
Drug: mFOLFOX6 — mFOLFOX6 administered as a combination of oxaliplatin and leucovorin as IV infusions. 5-FU administered as bolus followed by additional administration as IV infusion.
Drug: Placebo — IV infusion
  Arms: Placebo with mFOLFOX6

SUMMARY:
The main objective of this study is to compare efficacy of bemarituzumab combined with oxaliplatin, leucovorin, and 5-fluorouracil (5-FU) (mFOLFOX6) to placebo plus mFOLFOX6 as assessed by overall survival (OS) in participants with FGFR2b ≥10% 2+/3+ tumor cell staining (FGFR2b ≥10% 2+/3+TC)

ELIGIBILITY:
Inclusion Criteria:

* Adults with histologically documented unresectable, locally advanced or metastatic gastric or gastroesophageal junction cancer not amenable to curative therapy
* Fibroblast growth factor receptor 2b (FGFR2b) ≥10% 2+/3+ tumor cell staining as determined by centrally performed immunohistochemistry (IHC) testing, based on tumor sample either archival (obtained within 6 months/180 days prior to signing pre-screening informed consent) or a fresh biopsy
* Eastern Cooperative Oncology Group (ECOG) less than or equal to 1
* Measurable disease or non-measurable, but evaluable disease, according to Response Evaluation Criteria in Solid Tumors (RECIST) V 1.1
* Participant has no contraindications to mFOLFOX6 chemotherapy
* Adequate organ and bone marrow function:

  * absolute neutrophil count greater than or equal to 1.5 times 10^9/L
  * platelet count greater than or equal to 100 times 10^9/L
  * hemoglobin ≥ 9 g/dL without red blood cell (RBC) transfusion within 7 days prior to the first dose of study treatment
  * aspartate aminotransferase (AST) and alanine aminotransferase (ALT) less than 3 times the upper limit of normal (ULN) (or less than 5 times ULN if liver involvement). Total bilirubin less than 1.5 times ULN (or less than 2 times ULN if liver involvement); with the exception of participants with Gilbert's disease)
  * calculated or measured creatinine clearance (CrCl) of ≥ 30 mL/minute calculated using the formula of Cockcroft and Gault ([140 - Age]) × Mass [kg]/[72 × Creatinine mg/dL]) (x 0.85 if female)
  * international normalized ratio (INR) or prothrombin time (PT) less than 1.5 times ULN except for participants receiving anticoagulation, who must be on a stable dose of anticoagulant therapy for 6 weeks prior to enrollment

Exclusion Criteria:

* Prior treatment for metastatic or unresectable disease (Note: prior adjuvant, neo-adjuvant, and peri-operative therapy is allowed if completed more than 6 months prior to first dose of study treatment)
* Prior treatment with any selective inhibitor of fibroblast growth factor - fibroblast growth factor receptor (FGF-FGFR) pathway
* Known human epidermal growth factor receptor 2 (HER2) positive
* Untreated or symptomatic central nervous system (CNS) disease or brain metastases
* Peripheral sensory neuropathy greater than or equal to Grade 2
* Clinically significant cardiac disease
* Other malignancy within the last 2 years (exceptions for definitively treated disease)
* Chronic or systemic ophthalmological disorders
* Major surgery or other investigational study within 28 days prior to first dose of study treatment
* Palliative radiotherapy within 14 days prior to the first dose of study treatment
* Evidence of or recent history (within 6 months) of corneal defects, corneal ulcerations, keratitis, or keratoconus, history of corneal transplant, or other known abnormalities of the cornea that may pose an increased risk of developing a corneal ulcer.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 547 (Actual)
Dates: Start 2022-03-07 (Actual); Primary Completion 2025-06-20 (Actual); Study Completion 2026-06-20 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | Up to approximately 3.5 years
  Overall survival in FGFR2b ≥ 10% 2+/3+ tumor cell staining participants

SECONDARY OUTCOMES:
Progression-free Survival (PFS) | Up to approximately 3.5 years
  PFS in FGFR2b ≥ 10% 2+/3+ tumor cell staining participants
Objective Response Rate (ORR) | Up to approximately 3.5 years
  ORR in FGFR2b ≥ 10% 2+/3+ tumor cell staining participants
Number of Participants who Experience a Treatment-emergent Adverse Event (TEAE) | Up to approximately 3.5 years
  Any clinically significant changes in vital signs, visual acuity, and clinical laboratory tests after first dose will be recorded as TEAEs.
Overall Survival | Up to approximately 3.5 years
  Overall survival in all randomized participants
Progression-free Survival (PFS) | Up to approximately 3.5 years
  PFS in all randomized participants
Objective Response Rate (ORR) | Up to approximately 3.5 years
  ORR in all randomized participants
Duration of Response (DOR) | Up to approximately 3.5 years
  DOR in FGFR2b ≥ 10% 2+/3+ tumor cell staining participants
Disease Control Rate | Up to approximately 3.5 years
  Disease Control Rate in FGFR2b ≥ 10% 2+/3+ tumor cell staining participants
Mean Subjective Score in European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire (QLQ-C30) | Up to approximately 3.5 years
  Measured in FGFR2b ≥ 10% 2+/3+ tumor cell staining participants
Change from Baseline Score in European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire (QLQ-C30) | Baseline up to approximately 3.5 years
  Measured in FGFR2b ≥ 10% 2+/3+ tumor cell staining participants
Stomach Cancer Related Symptom Mean Subjective Score as Measured by European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire - Stomach (EORTC-QLQ-STO22) | Up to approximately 3.5 years
  Measured in FGFR2b ≥ 10% 2+/3+ tumor cell staining participants
Change from Baseline in Stomach Cancer Related Symptom Score as Measured by European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire - Stomach (EORTC-QLQ-STO22) | Baseline up to approximately 3.5 years
  Measured in FGFR2b ≥ 10% 2+/3+ tumor cell staining participants
Mean Subjective Score in Visual Analogue Scale (VAS) as Measured by the EuroQol 5-dimensional 5-levels (EQ-5D-5L) | Up to approximately 3.5 years
  Measured in FGFR2b ≥ 10% 2+/3+ tumor cell staining participants
Change from Baseline of Visual Analogue Scale (VAS) as Measured by the EuroQol 5-dimensional 5-levels (EQ-5D-5L) | Baseline up to approximately 3.5 years
  Measured in FGFR2b ≥ 10% 2+/3+ tumor cell staining participants
Time to Deterioration in Stomach Cancer Related Symptom Score as Measured by European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire - Stomach (EORTC-QLQ-STO22) | Up to approximately 3.5 years
  Measured in FGFR2b ≥ 10% 2+/3+ tumor cell staining participants
Time to Deterioration in European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire (QLQ-C30) Score | Up to approximately 3.5 years
  Measured in FGFR2b ≥ 10% 2+/3+ tumor cell staining participants
Time to Deterioration in Visual Analogue Scale (VAS) as Measured by the EuroQol 5-dimensional 5-levels (EQ-5D-5L) Score | Up to approximately 3.5 years
  Measured in FGFR2b ≥ 10% 2+/3+ tumor cell staining participants
Time to Deterioration in Physical Function Score as Measured by a Subscale of European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire (QLQ-C30) | Day 1 up to approximately 3.5 years
  Measured in FGFR2b ≥ 10% 2+/3+ tumor cell staining participants
Maximum Observed Concentration (Cmax) of Bemarituzumab in Combination with mFOLFOX6 in Plasma | Day 1 up to approximately 3.5 years
Observed Concentration at the End of a Dose Interval (Ctrough) of Bemarituzumab in Combination with mFOLFOX6 in Plasma | Day 1 up to approximately 3.5 years
Number of Participants with an Anti-bemarituzumab Antibody Formation | Day 1 up to approximately 3.5 years

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (299):
- United States (16):
  - Alaska Oncology and Hematology, Anchorage, Alaska
  - Mayo Clinic Arizona, Phoenix, Arizona
  - The Oncology Institute Clinical Research, Cerritos, California
  - University of California Los Angeles, Los Angeles, California
  - Mayo Clinic Florida, Jacksonville, Florida
  - Saint Francis Medical Group, Indianapolis, Indiana
  - University of Michigan, Ann Arbor, Michigan
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Healthier Hematology and Oncology Excelsior Integrated Medical Group, Brooklyn, New York
  - White Plains Hospital Center for Cancer Care, White Plains, New York
  - Levine Cancer Institute University, Charlotte, North Carolina
  - FirstHealth Cancer Center, Pinehurst, North Carolina
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Inova Schar Cancer Institute, Fairfax, Virginia
  - Medical Oncology Associates, PS, Spokane, Washington
- Argentina (8):
  - Instituto Alexander Fleming, CABA, Buenos Aires
  - Hospital Universitario Fundacion Favaloro, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - Sociedad de Beneficencia Hospital Italiano, Córdoba, Córdoba Province
  - Hospital Privado Universitario de Cordoba, Córdoba, Córdoba Province
  - Hospital Provincial del Centenario, Rosario, Santa Fe Province
  - Exelsus Oncologia Clinica, San Miguel de Tucumán, Tucumán Province
  - Instituto Argentino de Diagnostico y Tratamiento IADT, Buenos Aires
  - Hospital Britanico de Buenos Aires, Buenos Aires
- Australia (2):
  - Liverpool Hospital, Liverpool, New South Wales
  - St John of God Murdoch Hospital, Murdoch, Western Australia
- Belgium (4):
  - Universitair Ziekenhuis Antwerpen, Edegem
  - Universitair Ziekenhuis Gent, Ghent
  - Universitair Ziekenhuis Leuven - Campus Gasthuisberg, Leuven
  - Centre Hospitalier Universitaire de Liege - Sart Tilman, Liège
- Brazil (10):
  - Núcleo de Oncologia da Bahia, Salvador, Estado de Bahia
  - Centro de Oncologia Mackenzie, Curitiba, Paraná
  - Oncosite Centro de Pesquisa Clinica Em Oncologia Ltda, Ijuí, Rio Grande do Sul
  - Hospital Sao Lucas da Pontificia Universidade Catolica do Rio Grande do Sul, Porto Alegre, Rio Grande do Sul
  - Clinica de Oncologia Reichow, Blumenau, Santa Catarina
  - Centro de Pesquisa e Ensino em Oncologia de Santa Catarina, Florianópolis, Santa Catarina
  - Instituto de Ensino e Pesquisa Sao Lucas Iep Sao Lucas, Santo André, São Paulo
  - Instituto Nacional de Cancer, Rio de Janeiro
  - Hospital Nove de Julho - dasa, São Paulo
  - Instituto Brasileiro de Controle do Cancer Ibcc, São Paulo
- Bulgaria (6):
  - Multiprofile Hospital for Active Treatment Park Hospital EOOD, Branipole Village
  - Specialized Hospital for Active Treatment of Oncology - Haskovo EOOD, Haskovo
  - University Multiprofile Hospital for Active Treatment Dr Georgi Stranski EAD, Pleven
  - University Multiprofile Hospital for Active Treatment Pulmed OOD, Plovdiv
  - Acibadem City Clinic University Multiprofile Hospital for Active Treatment Tokuda EAD, Sofia
  - Multiprofile Hospital for Active Treatment Serdika EOOD, Sofia
- Canada (4):
  - Cross Cancer Institute, Edmonton, Alberta
  - The Ottawa Hospital Cancer Centre, Ottawa, Ontario
  - Sunnybrook Research Institute Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Jewish General Hospital, Montreal, Quebec
- Chile (4):
  - James Lind Centro de Investigacion del Cancer, Temuco, Cautín
  - Clinica CIDO, Temuco, Cautín
  - Centro de Estudios Clinicos SAGA Spa, Santiago
  - Centro de Estudios Clinicos e Investigaciones Medicas CeCim, Santiago
- China (59):
  - The First Affiliated Hospital of Bengbu Medical College, Bengbu, Anhui
  - The First Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - Anhui Provincial Cancer Hospital, Hefei, Anhui
  - Cancer Hospital of Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Chongqing University Three Gorges Hospital, Chongqing, Chongqing Municipality
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - The First Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - Lanzhou University Second Hospital, Lanzhou, Gansu
  - Gansu Wuwei Tumour Hospital, Wuwei, Gansu
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Guangdong Provincial Peoples Hospital, Guangzhou, Guangdong
  - Cancer Hospital of Shantou University Medical College, Shantou, Guangdong
  - The First Affiliated Hospital of Hainan Medical University, Haikou, Hainan
  - Fourth Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Tongji Hospital Affiliated to Tongji Medical College of Huazhong University of ScienceandTechnology, Wuhan, Hebei
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Anyang Cancer Hospital, Anyang, Henan
  - The First Affiliated Hospital of Henan University of science and Technology, Luoyang, Henan
  - Henan Cancer Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Taihe Hospital Affiliated Hospital of Hubei University of Medicine, Shiyan, Hubei
  - The Cancer Center Union Hospital Tongji Medical College Huazhong University of Science and Tech, Wuhan, Hubei
  - Hubei Cancer Hospital, Wuhan, Hubei
  - Xiangya Hospital of Central South University, Changsha, Hunan
  - Hunan Cancer Hospital, Changsha, Hunan
  - Nanjing First Hospital, Nanjing, Jiangsu
  - The Second Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - Affiliated Hospital of Jiangnan University, Wuxi, Jiangsu
  - The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The First Hospital of Jilin University, Changchun, Jilin
  - China-Japan Union Hospital of Jilin University, Changchun, Jilin
  - The First Affiliated Hospital of Jinzhou Medical University, Jinzhou, Liaoning
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - Liaoning Cancer Hospital, Shenyang, Liaoning
  - The First Affiliated Hospital of Xi an Jiaotong University, Xi'an, Shaanxi
  - Jinan Central Hospital, Jinan, Shandong
  - The Affiliated Cancer Hospital of Shandong First Medical University, Jinan, Shandong
  - The Affiliated Hospital of Qingdao University, Qingdao, Shandong
  - Zhongshan Hospital Fudan University, Shanghai, Shanghai Municipality
  - Shanghai General Hospital, Shanghai, Shanghai Municipality
  - Shanghai East Hospital, Shanghai, Shanghai Municipality
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Ruijin Hospital Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - Changzhi Peoples Hospital, Changzhi, Shanxi
  - Linfen Central Hospital, Linfen, Shanxi
  - Shanxi Province Cancer Hospital, Taiyuan, Shanxi
  - Sichuan Cancer Hospital, Chengdu, Sichuan
  - The First Affiliated Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - The Second Affiliated Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Sir Run Run Shaw Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Taizhou Hospital of Zhejiang Province, Linhai, Zhejiang
  - Lishui Municipal central Hospital, Lishui, Zhejiang
  - The First Affiliate Hospital of Ningbo University, Ningbo, Zhejiang
  - Peoples Hospital of Quzhou, Quzhou, Zhejiang
  - Beijing Cancer Hospital, Beijing
  - Tianjin Medical University Cancer institute and hospital, Tianjin
- Colombia (4):
  - Institucion Prestadora de Servicios de Salud Sociedad Médica Rionegro SA Somer SA, Rionegro, Antioquia
  - Sociedad de Oncologia y Hematologia del Cesar, Valledupar, Cesar Department
  - Fundacion Cardiovascular de Colombia, Bucaramanga, Santander Department
  - Instituto Cancerologico de Narino Ltda, Pasto
- Czechia (5):
  - Masarykuv onkologicky ustav, Brno
  - Fakultni nemocnice Hradec Kralove, Hradec Králové
  - Fakultni nemocnice Olomouc, Olomouc
  - Vseobecna fakultni nemocnice v Praze, Prague
  - Fakultni Thomayerova nemocnice, Prague
- Rigshospitalet, Copenhagen, Denmark
- North Estonia Medical Centre Foundation, Tallinn, Estonia
- France (13):
  - Centre Hospitalier Universitaire Amiens Picardie - Hopital Sud, Amiens
  - Sainte Catherine - Institut du Cancer d Avignon, Avignon
  - Centre Hospitalier Régional Universitaire de Besançon, Hôpital Jean Minjoz, Besançon
  - Centre Hospitalier Universitaire de Brest - Cavale Blanche, Brest
  - Centre Hospitalier Universitaire de Clermont Ferrand, Hôpital Estaing, Clermont-Ferrand
  - Centre Hospitalier Régional Universitaire de Lille - Hôpital Claude Huriez, Lille
  - Centre Leon Berard, Lyon
  - Hôpital Européen Georges Pompidou, Paris
  - Institut Mutualiste Montsouris, Paris
  - Centre Hospitalier Universitaire de Reims - Hôpital Robert Debré, Reims
  - Centre Hospitalier Universitaire Nord de Saint Etienne - Hôpital Nord, Saint-Priest-en-Jarez
  - Institut de cancerologie Strasbourg Europe, Strasbourg
  - Institut Gustave Roussy, Villejuif
- Greece (10):
  - Agios Savvas Anticancer Hospital, Athens
  - 251 General Airforce Hospital, Athens
  - General Hospital of Athens Laiko, Athens
  - Evgenidio Hospital I Agia Trias, Athens
  - Metropolitan Hospital, Athens
  - University Hospital of Heraklion, Heraklion - Crete
  - University Hospital of Larissa, Larissa
  - University Hospital of Patras, Pátrai
  - Anticancer Hospital of Thessaloniki Theageneio, Thessaloniki
  - Bioclinic of Thessaloniki, Thessaloniki
- Hungary (5):
  - Gyor-Moson-Sopron Varmegyei Petz Aladar Egyetemi Oktatokorhaz, Győr
  - Bekes Varmegyei Kozponti Korhaz Pandy Kalman Tagkorhaz, Gyula
  - Borsod-Abauj-Zemplen Varmegyei Kozponti Korhaz es Egyetemi Oktatokorhaz, Miskolc
  - Szabolcs-Szatmar-Bereg Varmegyei Oktatokorhaz Nyiregyhazi Josa Andras Tagkorhaz, Nyíregyháza
  - Tolna Varmegyei Balassa Janos Korhaz, Szekszárd
- Ireland (2):
  - St James Hospital, Dublin
  - St Vincents University Hospital, Dublin
- Israel (3):
  - Assuta Medical Center, Jerusalem
  - Hadassah Ein-Kerem Medical Center, Jerusalem
  - Meir Medical Center, Kfar Saba
- Italy (13):
  - Istituto Ospedaliero Fondazione Poliambulanza, Brescia
  - Azienda Ospedaliera di Rilievo Nazionale e Alta Specializzazione Garibaldi Nesima, Catania
  - Azienda Unita Sanitaria Locale LE Presidio Ospedaliero Vito Fazzi Polo Oncologico Giovanni Paolo II, Lecce
  - Azienda Socio Sanitaria Territoriale Grande Ospedale Metropolitano Niguarda, Milan
  - Azienda Ospedaliero Universitaria di Cagliari Policlinico Duilio Casula, Monserrato CA
  - Azienda Unita Saniataria Locale IRCCS di Reggio Emilia, Reggio Emilia
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Roma
  - Azienda Ospedaliera San Giovanni Addolorata, Roma
  - IRCCS Istituto Clinico Humanitas, Rozzano MI
  - Azienda Ospedaliera Ordine Mauriziano di Torino, Torino
  - Azienda Ospedaliera Cardinale Giovanni Panico, Tricase
  - Azienda Sanitaria Universitaria Friuli Centrale Presidio Ospedaliero Santa Maria della Misericordia, Udine
  - Azienda Ospedaliera Universitaria Integrata di Verona Ospedale Civile Maggiore Borgo Trento, Verona
- Japan (24):
  - Aichi Cancer Center, Nagoya, Aichi-ken
  - Nagoya University Hospital, Nagoya, Aichi-ken
  - Chiba Cancer Center, Chiba, Chiba
  - National Cancer Center Hospital East, Kashiwa-shi, Chiba
  - National Hospital Organization Shikoku Cancer Center, Matsuyama, Ehime
  - National Hospital Organization Kyushu Cancer Center, Fukuoka, Fukuoka
  - Gifu University Hospital, Gifu, Gifu
  - Hokkaido University Hospital, Sapporo, Hokkaido
  - Hyogo Cancer Center, Akashi-shi, Hyōgo
  - Kobe City Medical Center General Hospital, Kobe, Hyōgo
  - Ishikawa Prefectural Central Hospital, Kanazawa, Ishikawa-ken
  - Kagawa University Hospital, Kita-gun, Kagawa-ken
  - Yokohama City University Medical Center, Yokohama, Kanagawa
  - Kanagawa Prefectural Hospital Organization Kanagawa Cancer Center, Yokohama, Kanagawa
  - Kyoto University Hospital, Kyoto, Kyoto
  - Niigata Cancer Center Hospital, Niigata, Niigata
  - Kansai Medical University Hospital, Hirakata-shi, Osaka
  - Osaka International Cancer Institute, Osaka, Osaka
  - Kindai University Hospital, Osakasayama-shi, Osaka
  - Osaka University Hospital, Suita-shi, Osaka
  - Saitama Cancer Center, Kitaadachi-gun, Saitama
  - Shizuoka Cancer Center, Sunto-gun, Shizuoka
  - The Cancer Institute Hospital of Japanese Foundation for Cancer Research, Koto-ku, Tokyo
  - Keio University Hospital, Shinjuku-ku, Tokyo
- Pauls Stradins Clinical University Hospital, Riga, Latvia
- Lithuania (4):
  - Lietuvos sveikatos mokslu universiteto ligonine viesoji istaiga Kauno klinikos, Kaunas
  - Viesoji istaiga Klaipedos universitetine ligonine, Klaipėda
  - Nacionalinis vezio institutas, Vilnius
  - Vilnius University Hospital Santaros Clinic Public Institution, Vilnius
- Malaysia (3):
  - Hospital Kuala Lumpur, Kuala Lumpur, Kuala Lumpur
  - University Malaya Medical Centre, Kuala Lumpur, Kuala Lumpur
  - Sarawak General Hospital, Kuching, Sarawak
- Mexico (7):
  - Centro Oncologico Internacional, Tijuana, Baja California Norte
  - Hospital Civil de Guadalajara Fray Antonio Alcalde, Guadalajara, Jalisco
  - Investigacion Biomedica para el Desarrollo de Farmacos SA de CV, Zapopan, Jalisco
  - Christus Muguerza Clinica Vidriera, Monterrey, Nuevo León
  - Filios Alta Medicina sa de cv, Monterrey, Nuevo León
  - Investigación Biomédica para el Desarrollo de Fármacos, Aguascalientes
  - Trials In Medicine SC, México
- Oslo University Hospital, Oslo, Norway
- Peru (4):
  - Centro de Investigacion Clinica Trujillo Eirl, Trujillo, La Libertad
  - Instituto Peruano de Oncologia y Radioterapia, San Isidro, Lima region
  - Centro Medico Monte Carmelo, Arequipa
  - Oncosalud, Lima
- Poland (9):
  - Centrum Onkologii im prof Franciszka Lukaszczyka, Bydgoszcz
  - Szpitale Pomorskie Spzoo, Gdynia
  - Biokinetica SA, Józefów
  - Szpital Wojewodzki imienia Mikolaja Kopernika w Koszalinie, Koszalin
  - Szpital Kliniczny Ministerstwa Spraw Wewnetrznych i Administracji, Olsztyn
  - SPZOZ Opolskie Centrum Onkologii imienia prof Tadeusza Koszarowskiego w Opolu, Opole
  - Wielkopolskie Centrum Onkologii imienia Marii Sklodowskiej-Curie, Poznan
  - Wojewodzki Szpital im Sw Ojca Pio w Przemyslu, Przemyśl
  - Kliniki Neuroradiochirurgii Spzoo Radom Centr Onkolo im Bohater Radomsk Czerwca -76 Szpital Specjal, Radom
- Portugal (7):
  - Unidade Local de Saude de Coimbra, EPE, Coimbra
  - Unidade Local de Saude do Alto Ave, EPE, Guimarães
  - Unidade Local de Saude de Santa Maria, EPE - Hospital de Santa Maria, Lisbon
  - Unidade Local de Saude de Santo Antonio, EPE - Hospital de Santo Antonio, Porto
  - Instituto Portugues de Oncologia do Porto Francisco Gentil, EPE, Porto
  - Unidade Local de Saude de Sao Joao, EPE - Hospital de Sao Joao, Porto
  - Unidade Local de Saude de Entre Douro e Vouga, EPE - Hospital de Sao Sebastiao, Santa Maria da Feira
- Romania (6):
  - Spitalul Judetean de Urgenta Dr Constantin Opris Baia Mare, Baia Mare
  - Institutul Clinic Fundeni, Bucharest
  - Institutul Oncologic Prof Dr Alexandru Trestioreanu Bucuresti, Bucharest
  - SC Medisprof SRL, Cluj-Napoca
  - Institutul Regional de Oncologie Iasi, Iași
  - Ovidius Clinical Hospital, Ovidiu
- National Cancer Centre Singapore, Singapore, Singapore
- South Africa (4):
  - The Oncology Centre, Durban
  - Sandton Oncology Centre, Gauteng
  - Netcare Milpark Hospital, Johannesburg
  - Steve Biko Academic Hospital, Pretoria
- South Korea (15):
  - Dong-A University Hospital, Busan
  - Kyungpook National University Chilgok Hospital, Daegu
  - Chungnam National University Hospital, Daejeon
  - National Cancer Center, Goyang-si Gyeonggi-do
  - The Catholic University of Korea Incheon St Marys Hospital, Incheon
  - Jeonbuk National University Hospital, Jeonju-si, Jeollabuk-do
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Korea University Anam Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Kangbuk Samsung Hospital, Seoul
  - Severance Hospital Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - The Catholic University of Korea Seoul St Marys Hospital, Seoul
  - Korea University Guro Hospital, Seoul
- Spain (13):
  - Hospital Universitario Reina Sofia, Córdoba, Andalusia
  - Hospital Regional Universitario de Malaga, Málaga, Andalusia
  - Hospital Universitario Miguel Servet, Zaragoza, Aragon
  - Hospital Donostia, Donostia / San Sebastian, Basque Country
  - Hospital Universitario de Burgos, Burgos, Castille and León
  - Hospital Clinic i Provincial de Barcelona, Barcelona, Catalonia
  - Hospital de la Santa Creu i Sant Pau, Barcelona, Catalonia
  - Corporacio Sanitaria Parc Tauli, Sabadell, Catalonia
  - Complexo Hospitalario Universitario de Ourense, Ourense, Galicia
  - Hospital Universitari i Politecnic La Fe, Valencia, Valencia
  - Hospital General Universitario Gregorio Marañon, Madrid
  - Hospital Universitario Puerta de Hierro Majadahonda, Madrid
  - Hospital General Universitario Jose Maria Morales Meseguer, Murcia
- Sweden (3):
  - Sahlgrenska Universitetssjukhuset, Gothenburg
  - Karolinska Universitetssjukhuset Huddinge, Stockholm
  - Norrlands Universitetssjukhus, Umeå
- Taiwan (6):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - China Medical University Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - Tri-Service General Hospital, Taipei
  - Linkou Chang Gung Memorial Hospital of Chang Gung Medical Foundation, Taoyuan District
- Thailand (4):
  - King Chulalongkorn Memorial Hospital, Bangkok
  - Rajavithi Hospital, Bangkok
  - Ramathibodi Hospital, Bangkok
  - Siriraj Hospital, Bangkok
- Turkey (Türkiye) (17):
  - Baskent Universitesi Adana Doktor Turgut Noyan Uygulama ve Arastirma Merkezi, Adana
  - Doktor Abdurrahman Yurtaslan Ankara Onkoloji Egitim ve Arastirma Hastanesi, Ankara
  - Hacettepe Universitesi Tip Fakultesi Hastanesi, Ankara
  - Memorial Ankara Hastanesi, Ankara
  - Ankara Bilkent Sehir Hastanesi, Ankara
  - Antalya Egitim ve Arastirma Hastanesi, Antalya
  - Dicle Universitesi Tip Fakultesi, Diyarbakır
  - Bezmialem Vakif Universitesi Hastanesi, Istanbul
  - Istanbul Universitesi Cerrahpasa Tip Fakultesi, Istanbul
  - Goztepe Prof Dr Suleyman Yalcin Sehir Hastanesi, Istanbul
  - Kartal Dr Lutfi Kirdar Sehir Hastanesi, Istanbul
  - Izmir Ataturk Egitim ve Arastirma Hastanesi, Izmir
  - Kocaeli Universitesi Tip Fakultesi Hastanesi, Kocaeli
  - Inonu Universitesi Turgut Ozal Tip Merkezi, Malatya
  - Sakarya Egitim ve Arastirma Hastanesi, Sakarya
  - Ondokuz Mayis Universitesi Tip Fakultesi Hastanesi, Samsun
  - Van Yuzuncu Yil Universitesi Dursun Odabas Tip Merkezi, Van

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: https://www.amgen.com/datasharing

REFERENCES:
- [Background] Rha SY, Zhang Y, Elme A, Pazo Cid R, Alacacioglu A, Ziogas DC, Shitara K, Ranceva A, Nemecek R, Santoro A, Calderon CA, Korphaisarn K, Davis T, Zahlten-Kuemeli A, Conn C, Tan M, Honeycutt H, Wainberg ZA. Prevalence of FGFR2b Protein Overexpression in Advanced Gastric Cancers During Prescreening for the Phase III FORTITUDE-101 Trial. JCO Precis Oncol. 2025 Jan;9:e2400710. doi: 10.1200/PO-24-00710. Epub 2025 Jan 24. PMID 39854659
- [Background] Farooq AV, Kaur S, Hundal P, Burke M, Sulaiman R, Zahlten-Kumeli A, Raoof S, Li Z, Murias Dos Santos T, Huang XJ, Colby K. Advancing Ocular Safety Profile Assessment: A Novel Grading Scale for Ocular Adverse Reactions Associated with Bemarituzumab. Ophthalmol Ther. 2025 Jul;14(7):1349-1356. doi: 10.1007/s40123-025-01139-6. Epub 2025 May 12. PMID 40355729
- [Derived] Wainberg ZA, Kang YK, Lee KW, Qin S, Yamaguchi K, Kim IH, Saeed A, Oh SC, Li J, Turk HM, Teixeira A, Hitre E, Udrea AA, Cardellino GG, Sanchez RG, Zahlten-Kumeli A, Taylor K, Enzinger PC. Bemarituzumab as first-line treatment for locally advanced or metastatic gastric/gastroesophageal junction adenocarcinoma: final analysis of the randomized phase 2 FIGHT trial. Gastric Cancer. 2024 May;27(3):558-570. doi: 10.1007/s10120-024-01466-w. Epub 2024 Feb 3. PMID 38308771
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com